CLINICAL TRIAL: NCT02065856
Title: An Open Trial to Assess the Tolerability of AVANZ® Salsola Immunotherapy
Acronym: AV-X-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013-001728-20; 2013-001728-20 (EudraCT Number)
Record Dates: First submitted 2014-01-20; First posted 2014-02-19 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Allergic Rhinoconjunctivitis Due to Salsola Kali Pollen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVANZ Salsola kali (Experimental): Subcutaneous immunotherapy
  Interventions: Biological: AVANZ Salsola

INTERVENTIONS:
Biological: AVANZ Salsola — AVANZ Salsola

SUMMARY:
This trial is an open, national, multi-centre trial. The trial will be initiated in December 2013 and subjects will receive treatment for 6 weeks.

Safety monitoring will be performed in an ongoing basis through a Clinical Safety Group with immediate access to Adverse Events registered in the clinical database. The composition, procedures and deliverables of the Clinical Safety Group will be detailed in a Safety Agreement prior to trial start.

ELIGIBILITY:
Inclusion Criteria:

* A clinical history of Salsola kali pollen induced allergic rhinoconjunctivitis with or without asthma at least one year prior to trial entry.
* Positive Skin Prick Test to Salsola kali pollen (wheal diameter ≥ 3 mm).
* Documenting in the last 5 years a positive specific Immunoglobulin E against Salsola kali pollen (≥ Class 2; ≥0.70 KU/L).

Exclusion Criteria:

* Forced expiratory volume at one second 1 < 70% of predicted value at screening after adequate pharmacologic treatment.
* Uncontrolled or severe asthma.
* History of severe asthma exacerbation or emergency room visit or admission for asthma in the previous 12 months.
* At screening, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infection (serous otitis media is not an exclusion criterion).
* Treatment with parenteral corticosteroids, oral corticosteroids or anti-IgE in the previous 3 months or during the study (except for steroids if needed as rescue medication).
* Currently treated with angiotensin converting enzyme (ACE) inhibitors, tricyclic antidepressants, β-blockers, mono amine oxidase inhibitors (MAOIs) and any other drug containing alum (e.g. antacids) taken on a daily basis.
* Immunotherapy with Cupressus arizonica or Salsola kali pollen extracts within the previous 5 years (initiation of subcutaneous immunotherapy is acceptable if treatment has been discontinued before reaching maintenance dose; for SLIT 3 months in the last 5 years is accepted) or concomitant immunotherapy with any other allergen.
* History of anaphylactic shock due to e.g. food, insect venom, exercise or drug.
* History of severe and recurrent angioedema.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with adverse reactions | Participants will be followed for an expected average of 6 weeks

SECONDARY OUTCOMES:
Frequency of patients with systemic reactions according to EAACI classification | Participants will be followed for an expected average of 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: PURIFICACION GONZÁLEZ, PhD, Principal Investigator — Hospital General Universitario de Alicante
Locations (1):
- Hospital General Universitario de Alicante, Alicante, Alicante, Spain